CLINICAL TRIAL: NCT01463046
Title: A Phase I Dose Finding and Proof-of-concept Study of the Histone Deacetylase Inhibitor Panobinostat (LBH589) in Combination With Standard Dose Cytarabine and Daunorubicin for Older Patients With Untreated Acute Myeloid Leukemia or Advanced Myelodysplastic Syndrome
Brief Title: Phase I Dose Finding and Proof-of-concept Study of Panobinostat With Standard Dose Cytarabine and Daunorubicin for Untreated Acute Myeloid Leukemia or Advanced Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112512
Record Dates: First submitted 2011-10-27; First posted 2011-11-01 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Acute Myeloid Leukemia; Advanced Myelodysplastic Syndrome
Keywords: leukemia; AML; AMS; panobinostat; cytarabine; daunorubicin; HDAC
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Panobinostat; Cytarabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Panobinostat (Experimental)
  Interventions: Drug: Panobinostat; Drug: Cytarabine; Drug: Daunorubicin

INTERVENTIONS:
Drug: Panobinostat — Induction - 20-60 mg (1-3 20 mg capsules) PO on days 1,3,5 and 8
  Second induction - 20-60 mg (1-3 20 mg capsules) PO days 1,3 and 5
  Consolidation - 20-60 mg (1-3 20 mg capsules) PO on days 1,3,5 and 8
  Other Names: LBH589
Drug: Cytarabine — Induction - 100 mg/m2 continuous IV daily for 7 doses on day 3-9.
  Second induction - 100 mg/m2 continuous IV daily for 7 doses on day 3-7.
  Dosing for consolidation - 100 mg/m2 continuous IV daily for 7 doses on day 3-9.
  Other Names: ara-C
Drug: Daunorubicin — Induction - 60 mg/m2 IV over 15-30 minutes daily for 3 doses on day 3-5.
  Second induction - 60 mg/m2 IV over 15-30 minutes daily for 2 doses on day 3 and 4.
  Dosing for consolidation - 60 mg/m2 IV over 15-30 minutes daily for 3 doses on day 3-5.
  Other Names: Cerubidine

SUMMARY:
The purpose of this study is to see if Panobinostat is safe to give to patients and to determine the best dose to give in combination with standard cytarabine and daunorubicin chemotherapy.

DETAILED DESCRIPTION:
In the United States, the incidence of acute myeloid leukemia (AML) is approximately 3.5 cases per 100,000 persons per year. Approximately 13,000 people were diagnosed with AML in 2009 and 9,000 died of the disease, making AML the 6th leading cause of cancer death. Over the past three decades, AML survival has improved for younger patients with 5-year survival rates of greater than 60% for adults under the age of 45 years likely owing to improvements in induction and consolidation chemotherapy, allogeneic hematopoietic stem cell transplant (HSCT) and supportive care. Post-remission therapy with high-dose cytarabine-based regimens after cytarabine and anthracycline based induction has improved disease free and overall survival at the expense of increased treatment related mortality limiting its use in many older patients and those with significant comorbidities. Although allogeneic HSCT remains the standard of care for patients with poor risk AML or relapsed disease, advanced age, comorbidities and donor availability preclude this option for a large number of patients making improvement in the tolerability and efficacy of induction therapy an important goal.

Over half of newly diagnosed AML patients are over 65 years of age with a third over the age of 75 years. Unlike younger patients, the prognosis of elderly patients with AML is still dismal with five-year survival rates of less than 10% for patients over the age of 65 years. For the last thirty years, induction therapy with standard dose cytarabine with an anthracycline has remained the standard of care for elderly patients with AML. In the elderly, complete response rates to induction chemotherapy are lower than younger patients at 40 to 60% with median survival approaching 12 months. New strategies using novel agents to increase the sensitivity of malignant myeloid precursors to standard induction chemotherapy may improve complete response and relapse rates without increasing treatment related mortality.

Myelodysplastic syndromes (MDS)

The myelodysplastic syndromes are neoplasms of hematopoietic progenitor cells characterized by ineffective hematopoiesis and increased risk of transformation to AML. Clinically, patients develop symptoms related to with cytopenias, typically progressive anemia with or without thrombocytopenia or neutropenia that is unrelated to a defined reversible cause such as nutritional deficiency. Histologically, MDS is suggested by the presence of dysplasia in >10% of cells in one or more myeloid lineage on bone marrow evaluation. Characteristic cytogenetic abnormalities also aid in making the diagnosis of MDS.

The incidence of MDS in the U.S. has been estimated at 3.4 cases per 100,000 people per year with the incidence increasing 10 fold in people over the age of 70. Risk factors for the development of MDS include advanced age, male sex, and prior exposure to DNA-damaging chemotherapy or radiation therapy, typically for treatment of other malignancies. As a group, patients with advanced MDS and those with MDS progressing to AML have treatment resistant disease with low response rates and short durations of response after induction therapy.

The International Prognostic Scoring System (IPSS) for primary MDS assigns four MDS risk categories (Low, INT-1, INT-2, High) based on bone marrow myeloblast percentage, specific cytogenetic abnormalities, and number of cytopenias to estimate survival and risk of transformation to AML. Low and INT-1 risk MDS patients have a median survival of 5.7 and 3.3 years, respectively, in the absence of therapy. Advanced MDS patients in IPSS risk groups INT-2 and High fare much less well with median survival of 1.1 and 0.4 years, respectively. INT-2 and High-risk MDS is also associated with a higher risk of transformation to AML. In addition, hematopoietic precursors from patients with advanced MDS more frequently express the multi-drug resistance (MDR1) gene product P-glycoprotein, possibly explaining the low response rates and short duration of responses in this group after conventional induction therapies. A Phase III trial of the P-glycoprotein inhibitor valspodar in combination with mitoxantrone, etoposide and cytarabine in relapsed or refractory AML and high-risk MDS failed to show improved outcomes with P-glycoprotein inhibition. As such, novel therapeutic strategies to overcome the intrinsic resistance to chemotherapy seen in advanced MDS are needed to improve induction chemotherapy as primary therapy and as a bridge to allogeneic hematopoietic cell transplant.

Given the relatively long survival and low rate of progression to AML seen in patients with IPSS Low and INT-1 risk disease, allogeneic transplant is typically reserved for those who fail conservative management with erythropoiesis stimulating agents, G-CSF, hypomethylating agents such as azacitidine or decitabine, lenalidomide, or immune suppression therapy. For patients 60 years of age and younger with advanced MDS (INT-2, High), allogeneic hematopoietic cell transplant is the most appropriate therapy as it prolongs life expectancy. Due to advanced age and significant co-morbidities, allogeneic hematopoietic transplant is not an appropriate treatment modality for a large number of patients with advanced MDS. In addition, stem cell donors are not available for all patients. For patients with advanced MDS, hypomethylating agents or enrollment on clinical trials are both appropriate treatment options given the poor outcomes in this patient population. A phase III open-label, randomized trial of azacitidine versus conventional care regimens in advanced MDS showed superior overall survival for patients treated with azacitidine (24.5 versus 15.0 months, HR 0.58; 95% CI 0.43-0.77). Although decitabine has activity in MDS, it has not been shown to prolong survival in advanced MDS to date. In a phase III study comparing decitabine to supportive care, decitabine showed a superior response rate and delayed the time to the development of AML.

Anthracyclines in AML therapy

Anthracycline chemotherapy agents (daunorubicin, idarubicin, mitoxantrone) are highly active in AML and are an essential part initial induction therapy in those fit for intensive chemotherapy. The optimal dose of anthracycline to maximize response and survival while preserving safety is still being determined. For daunorubicin, a Phase III randomized study of younger patients ages 17 to 60 years with AML demonstrated that standard dose cytarabine 100 mg/m2 daily for 7 days in combination with daunorubicin 90 mg/m2 daily for 3 days was superior to daunorubicin 45 mg/m2 daily for 3 days with improved complete remission rates (70.6% vs. 57.3%, p<0.001) and median overall survival (23.7 vs. 15.7 months, p=0.003). Toxicity was not significantly different between the two groups. A similar Phase III study in AML patients 60 years of age or older compared daunorubicin 45 mg/m2 to 90 mg/m2 for 3 days in combination with cytarabine 200 mg/m2 daily for 7 days. Although the complete remission rate was higher in patients receiving the 90 mg/m2 daunorubicin dose (64% vs 54%, p=0.002), no difference was seen in survival. Notably, patients aged 60-65 years receiving higher daunorubicin dose had superior complete remission rates, event-free survival and overall survival. To date, no head-to-head comparisons of daunorubicin at 60 mg/m2 versus 90 mg/m2 have been published.

Histone deacetylases and their inhibitors in AML and MDS

HDAC inhibitors have shown activity in Phase I monotherapy trials for AML and advanced MDS. A Phase I trial of panobinostat as monotherapy in primarily AML yielded transient hematologic responses with reduction in peripheral blood blast counts in 8 of 11 patients consistent with the documented in vitro activity of the drug. Major toxicities included nausea, diarrhea, hypokalemia, anorexia, thrombocytopenia and reversible QTcF prolongation. Similar responses with rare complete responses have also been seen with the HDAC inhibitors romidepsin and MGCD0103 in AML and MDS.

Synergy between HDAC inhibitors and anthracyclines

As monotherapy, HDAC inhibitors are unlikely to impact the treatment of AML and advanced MDS although there is a strong biologic rationale for use of these agents in combination therapies. By inhibiting deacetylation of histones, HDAC inhibitors generate a more open chromatin structure more susceptible to the DNA damaging effects of anthracycline chemotherapeutic agents, in some instances when administered 48 hours after the HDAC inhibitor. In vitro, HDAC inhibitors potentiate the cytotoxic effects of anthracyclines in leukemia cell lines. Panobinostat, specifically, acts synergistically with the anthracycline doxorubicin to induce DNA damage, increase histone acetylation and activate programmed cell death in AML cell lines and primary AML cells. The administration of the anthracycline daunorubicin with panobinostat is predicted to be synergistic in vivo and may improve complete response and relapse rates for AML.

Proper sequencing of HDAC inhibitors with anthracyclines will likely be important to the success of these combinations. Pretreatment with HDAC inhibitors prior to anthracycline exposure may provide synergistic effects as well by increasing nuclear DNA exposure to anthracycline. In cultured MCF-7 breast cancer cells, treatment with the HDAC inhibitor vorinostat leads to chromatin decondensation which is maximal after 48 hours of HDAC inhibitor treatment. In this system, co-administration of vorinostat and epirubicin did not lead to increased apoptosis whereas 48 hour pre-incubation with vorinostat led to synergistic increases in apoptosis associated with increased nuclear accumulation of epirubicin and increased DNA damage. In AML, maximal epigenetic effects appear to occur at about 48 hours after HDAC inhibitor exposure as well.

Anticancer activity of DAC inhibitors

Alterations in chromosome structure play critical roles in the control of gene transcription. These epigenetic alterations include modification of histones and others proteins by acetylation and/or phosphorylation. Normally, these modifications are balanced finely and are highly reversible in normal tissues, but they may be imbalanced and heritable in tumor cells. DAC inhibitors increase histone acetylation, thereby modulating the expression of a subset of genes in a coordinated fashion. Several tumors suppressor genes associated with the malignant phenotype are repressed by epigenetic mechanisms in sporadic cancers. Thus therapy with DAC inhibitors may alter tumor phenotype and inhibit growth in such tumors.

Multiple hallmarks of cancer are regulated by acetylation/deacetylation:

* DAC inhibition targets both histone and nonhistone proteins. Targeting the acetylation status of nonhistone, tumor-associated proteins that mediate proliferation may be the underlying antitumor mechanism of DAC inhibitors.
* Nonhistone proteins regulated by acetylation include α-tubulin, p53, HIF-1α, and HSP90. These proteins are substrates of DACs.
* The ability of a single agent to target multiple molecular features of tumor cells may result in good efficacy against a range of different tumor types.
* HSP90 is involved in protein stability and degradation; the inhibition of HSP90 affects protein turnover in diseases such as multiple myeloma and B-cell malignancies.
* Acetylated HIF-1α is degraded and can no longer act as a tumor growth factor. Class II DAC inhibitors target histone deacetylase (HDAC or DAC) 6, resulting in increased acetylation of HIF-1α and decreased vascular endothelial growth factor (VEGF), thereby inhibiting angiogenesis.
* Both acetylation and ubiquitylation often occur on the same lysine residue, but these processes cannot occur simultaneously. Acetylation allows for increased stability, and ubiquitylation leads to protein degradation. Therefore, DACs decrease the half-life of a protein by exposing the lysine residue for ubiquitylation.

Panobinostat (LBH589)

Panobinostat (LBH589) is a deacetylase inhibitor (DACi) belonging to a structurally novel cinnamic hydroxamic acid class of compounds. It is a potent class I/II pan-DAC inhibitor (pan-DACi) that has shown anti-tumor activity in pre-clinical models and cancer patients. Deacetylases (DAC) target lysine groups on chromatin and transcription factors and various non-histone proteins such as p53, tubulin, HSP90 and Rb. Panobinostat is formulated as an oral capsule and a solution for intravenous (i.v.) injection. Both the oral and i.v. formulations are currently being investigated in ongoing Phase I and Phase II studies in advanced solid tumors and hematological malignancies.

Inhibition of DAC provides a novel approach for cancer treatment. Histones are part of the core proteins of nucleosomes, and acetylation and deacetylation of these proteins play a role in the regulation of gene expression. Highly charged deacetylated histones bind tightly to the phosphate backbone of DNA, inhibiting transcription, presumably, by limiting access of transcription factors and RNA polymerases to DNA. Acetylation neutralizes the charge of histones and generates a more open DNA conformation. This conformation allows transcription factors and associated transcription apparatus access to the DNA, promoting expression of the corresponding genes. The opposing activities of two groups of enzymes, histone acetyltransferase (HAT) and DAC control the amount of acetylation. In normal cells a balance exists between HAT and DAC activity that leads to cell specific patterns of gene expression. Perturbation of the balance produces changes in gene expression.

Several lines of evidence suggest that aberrant recruitment of DAC and the resulting modification of chromatin structure may play a role in changing the gene expression seen in transformed cells. For example, silencing of tumor suppressor genes at the level of chromatin is common in human tumors and DAC complexes have been shown to be crucial to the activity of the AML-specific fusion proteins PLZF-RAR-α, PML-RAR-α, and AML1/ETO. DAC inhibitors (DACi) have been shown to induce differentiation, cell cycle arrest or apoptosis in cultured tumor cells, and to inhibit the growth of tumors in animal models. In addition, DACi have been shown to induce expression of p21, a key mediator of cell cycle arrest in G1 phase and cellular differentiation.

Tumor growth inhibition and apoptosis in response to DACi treatment may also be mediated through changes in acetylation of non-histone proteins (e.g., HSP90, p53, HIF-1α, α-tubulin). For example, the chaperone protein HSP90 has been shown to be acetylated in cells treated with DACi. Acetylation of HSP90 inhibits its ability to bind newly synthesized client proteins, thus preventing proper client protein folding and function. In the absence of HSP90 function, misfolded proteins are targeted for degradation in the proteasome. Many proteins that require HSP90 association are critical to cancer cell growth, including ErbB1, ErbB2, AKT, Raf, KDR, and BCR-ABL. Acetylation of HSP90 in cells treated with DACi inhibits the chaperone function of HSP90, leading to degradation of the client proteins and eventual cell death.

The potential clinical utility of the use of DACi in cancer therapy was first suggested by the activity of the DACi, sodium phenylbutyrate, against acute promyelocytic leukemia (APL). An adolescent female patient with relapsed APL, who no longer responded to all trans-retinoic acid (ATRA) alone, achieved a complete clinical remission after treatment with a combination of ATRA and the DACi sodium phenylbutyrate.

ELIGIBILITY:
Inclusion Criteria:

* Untreated histologically confirmed acute myeloid leukemia OR advanced myelodysplastic syndrome (INT-2 or High risk) not previously treated with anthracycline-based chemotherapy OR a therapy-related myeloid neoplasm
* Male or female aged ≥ 60 years
* ECOG performance status 0-2
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Absence of major metabolic, renal and hepatic impairment as defined by the following laboratory parameters: AST and ALT ≤ 2.5 x ULN Serum bilirubin ≤ 1.5 x ULN Albumin > 3.0 g/dl Serum potassium ≥ LLN Total serum calcium [corrected for serum albumin] or ionized calcium ≥LLN Serum magnesium ≥ LLN
* Clinically euthyroid. Note: Patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism.
* Prior treatment of myelodysplastic syndrome or myeloproliferative neoplasm acceptable

Exclusion Criteria:

* Acute promyelocytic leukemia (FAB M3 AML)
* Known central nervous system involvement by leukemia
* Isolated myeloid sarcoma not meeting bone marrow criteria for AML or MDS
* Cumulative anthracycline exposure greater than 200 mg/m2 doxorubicin isotoxic equivalents (See Appendix A6 for conversions)
* Prior HDAC inhibitor, DAC inhibitor, Hsp90 inhibitor or valproic acid for the treatment of cancer
* Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first panobinostat treatment
* Prior allogeneic hematopoietic stem cell transplant
* Prior solid organ transplant
* Active bleeding diathesis or current treatment with therapeutic doses of sodium warfarin (Coumadin®) or other vitamin K active agents (Note: mini-dose of Coumadin® (e.g., 1 mg/day) or anti-coagulants given to maintain intravenous line patency, as well as unfractionated or low molecular weight heparin therapy are permitted)
* Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

History or presence of sustained ventricular tachyarrhythmia. (Patients with a history of atrial arrhythmia are eligible but should be discussed with Novartis prior to enrollment) Any history of ventricular fibrillation or torsade de pointes Bradycardia defined as HR< 50 bpm. Patients with pacemakers are eligible if HR ≥ 50 bpm Screening ECG with a QTcF > 450 msec Right bundle branch block + left anterior hemiblock (bifascicular block) Patients with myocardial infarction or unstable angina ≤ 6 months prior to starting study drug Congestive heart failure (CHF) that meets New York Heart Association (NYHA) Class II to IV definitions and/or ejection fraction <50% by MUGA scan or by transthoracic echocardiogram Other clinically significant heart disease (e.g. uncontrolled hypertension, or history of labile hypertension)

* Impairment of GI function or GI disease that may significantly alter the absorption of panobinostat.
* Patients with active diarrhea > CTCAE grade 2
* Known HIV infection
* Known active Hepatitis B or Hepatitis C virus infection
* Other concurrent severe and/or uncontrolled medical conditions (e.g. uncontrolled diabetes or active or uncontrolled infection) including abnormal laboratory values that could in the opinion of the investigator cause unacceptable safety risks or compromise compliance with the protocol.
* Active second malignancy except localized prostate cancer, basal cell carcinoma of the skin and carcinoma in situ of the skin or cervix
* Patients who are unwilling to stop the use of herbal remedies while on the Treatment Phase of the study
* Concomitant use of drugs with a risk of prolonging the QT interval and/or causing torsades de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug. Concomitant use of strong CYP3A4 inhibitors.
* Patients who have received targeted agents within 2 weeks or within 5 half-lives of the agent and active metabolites (which ever is longer) and who have not recovered from side effects of those therapies.
* Patients who have received either immunotherapy within < 8 weeks; chemotherapy within < 4 weeks; or radiation therapy to > 30% of marrow-bearing bone within < 2 weeks prior to starting study treatment; or who have not yet recovered from side effects of such therapies.
* Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Treatment with investigational agent within 30 days prior to enrollment
* Male patients whose sexual partners are women of childbearing potential not using a double method of contraception during the study and 3 months after the end of treatment. One of these methods must be a condom.
* Unwilling to accept blood product transfusions
* Unable to swallow pills
* Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-01; Primary Completion 2015-11-14 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) for the combination of panobinostat with standard-dose cytarabine and daunorubicin (7+3) for untreated AML and advanced MDS in the elderly. | Start of induction therapy until 21 days after the last dose of induction or second induction therapy or until count recovery in patients without residual disease, whichever is longer
The recommended Phase II dose for the combination of panobinostat with standard-dose cytarabine and daunorubicin (7+3) for untreated AML and advanced MDS in the elderly. | Start of induction therapy until 21 days after the last dose of induction or second induction therapy or until count recovery in patients without residual disease, whichever is longer

SECONDARY OUTCOMES:
Response rate (OR, CR, CRi) for AML using Revised Recommendations of the International Working Group | 18 days after the start of induction therapy or 37 days after the second induction therapy or when white blood cell count recovers, whichever is first.
Response rate (OR, CR, CRi) for AMS using International Working Group response criteria in myelodysplasia | 18 days after the start of induction therapy or 37 days after the second induction therapy or when white blood cell count recovers, whichever is first.
Relapse-free survival | The time to relapse or death from any cause from the date of confirmed morphologic CR.
Overall Survival | The time to death from any cause from the day 1 of induction therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Charalambos Andreadis, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States